CLINICAL TRIAL: NCT01750086
Title: Acute Effect of Teriparatide With Bisphosphonate or Denosumab on Bone Resorption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001956
Record Dates: First submitted 2012-11-26; First posted 2012-12-17 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: osteoporosis; postmenopausal; denosumab; teriparatide; alendronate; Forteo®; Prolia®
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide; Injections, Subcutaneous; Denosumab; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab 60mg subcutaneous injection (Active Comparator): Each subject will receive one teriparatide 40-mcg subcutaneous injection at each study visit.
  Interventions: Drug: Teriparatide 40-mcg subcutaneous injection; Drug: Denosumab Injection
- Alendronate 70mg weekly x 8 weeks (Active Comparator): Each subject will receive one teriparatide 40-mcg subcutaneous injection at each study visit.
  Interventions: Drug: Teriparatide 40-mcg subcutaneous injection; Drug: Alendronate Oral Tablet

INTERVENTIONS:
Drug: Teriparatide 40-mcg subcutaneous injection
  Other Names: Forteo®
Drug: Denosumab Injection — One-time Denosumab injection
  Arms: Denosumab 60mg subcutaneous injection
Drug: Alendronate Oral Tablet — weekly alendronate for 8 weeks
  Arms: Alendronate 70mg weekly x 8 weeks

SUMMARY:
The aim of the study is to assess the relative antiresorptive properties of 2 osteoporosis medications when combined with teriparatide.

ELIGIBILITY:
Inclusion Criteria:

Must satisfy A and B and C below:

A. Women aged 45+

B. Postmenopausal

C. Osteoporotic with high risk of fracture

Exclusion Criteria:

* History of significant hepatic, renal, cardiovascular, malignant disease, or conditions with impaired immune system
* Current alcohol or substance abuse
* Major psychiatric disorders
* Abnormal calcium level, elevated PTH, vitamin D deficiency, or anemia
* Known congenital or acquired bone disease other than osteoporosis
* Current use or past use in the past 12 months of oral bisphosphonates
* Current use or use in the past 3 months of estrogens, selective estrogen receptor modulators, or calcitonin
* Use of oral or parenteral glucocorticoids for more than 14 days in the past 6 months
* Any current or previous use of strontium or intravenous bisphosphonates
* Sensitivity to cell-derived drug products or teriparatide
* Extensive dental work involving dental extraction or dental implant within the past 2 months or in the upcoming 2 months
* Inability to sit upright for 30 minutes
* Esophageal abnormalities

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Cosman F, Eriksen EF, Recknor C, Miller PD, Guanabens N, Kasperk C, Papanastasiou P, Readie A, Rao H, Gasser JA, Bucci-Rechtweg C, Boonen S. Effects of intravenous zoledronic acid plus subcutaneous teriparatide [rhPTH(1-34)] in postmenopausal osteoporosis. J Bone Miner Res. 2011 Mar;26(3):503-11. doi: 10.1002/jbmr.238. PMID 20814967
- [Background] Finkelstein JS, Hayes A, Hunzelman JL, Wyland JJ, Lee H, Neer RM. The effects of parathyroid hormone, alendronate, or both in men with osteoporosis. N Engl J Med. 2003 Sep 25;349(13):1216-26. doi: 10.1056/NEJMoa035725. Epub 2003 Sep 20. PMID 14500805
- [Background] Cosman F, Nieves J, Zion M, Woelfert L, Luckey M, Lindsay R. Daily and cyclic parathyroid hormone in women receiving alendronate. N Engl J Med. 2005 Aug 11;353(6):566-75. doi: 10.1056/NEJMoa050157. PMID 16093465
- [Background] Kostenuik PJ, Capparelli C, Morony S, Adamu S, Shimamoto G, Shen V, Lacey DL, Dunstan CR. OPG and PTH-(1-34) have additive effects on bone density and mechanical strength in osteopenic ovariectomized rats. Endocrinology. 2001 Oct;142(10):4295-304. doi: 10.1210/endo.142.10.8437. PMID 11564687
- [Background] Finkelstein JS, Wyland JJ, Lee H, Neer RM. Effects of teriparatide, alendronate, or both in women with postmenopausal osteoporosis. J Clin Endocrinol Metab. 2010 Apr;95(4):1838-45. doi: 10.1210/jc.2009-1703. Epub 2010 Feb 17. PMID 20164296
- [Derived] Tsai JN, Zhu Y, Foley K, Lee H, Burnett-Bowie SA, Neer RM, Leder BZ. Comparative Resistance to Teriparatide-Induced Bone Resorption With Denosumab or Alendronate. J Clin Endocrinol Metab. 2015 Jul;100(7):2718-23. doi: 10.1210/jc.2015-1541. Epub 2015 May 1. PMID 25933031

RESULTS

PARTICIPANT FLOW:
Groups:
- Denosumab 60mg Subcutaneous Injection; Alendronate 70mg Weekly x 8 Weeks: Each subject will receive one teriparatide 40-mcg subcutaneous injection at each study visit.
  Teriparatide 40-mcg subcutaneous injection
Period: Overall Study
Arm/Group | Denosumab 60mg Subcutaneous Injection | Alendronate 70mg Weekly x 8 Weeks
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60mg Subcutaneous Injection | Alendronate 70mg Weekly x 8 Weeks | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7) | 66 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Bone Turnover Marker (Blood Sample)
Description: The primary outcome was the between-group difference in the teriparatide-induced change in serum c-telopeptide from baseline to week 8.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in CTX
Arm/Group | Denosumab 60mg Subcutaneous Injection | Alendronate 70mg Weekly x 8 Weeks
Number analyzed (Participants) | 12 | 13
percentage of change in CTX | -7 (11) | 43 (29)

ADVERSE EVENTS:
Arm/Group | Denosumab 60mg Subcutaneous Injection | Alendronate 70mg Weekly x 8 Weeks
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 60mg Subcutaneous Injection (N=12) | Alendronate 70mg Weekly x 8 Weeks (N=13)
Lightheadedness (Endocrine disorders) | 1 | 0 — One subject experienced lightheadedness 3 hours after the first teriparatide injection
Syncope (Endocrine disorders) | 0 | 1 — One subject experienced lightheadedness and syncope 3 hours after the first teriparatide injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No